CLINICAL TRIAL: NCT01318889
Title: Effects of Topical Dexpanthenol on Chemotherapy and Radiotherapy Induced Oral Mucositis
Brief Title: Dexpanthenol Mouthwash to Treat Oral Mucositis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Dr Anbari, Dental Faculty of shaheed Beheshti medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMU1360
Record Dates: First submitted 2011-03-08; First posted 2011-03-21 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2010-06

CONDITIONS: Oral Mucositis (Ulcerative) Due to Radiation
Keywords: Dexpanthenol; Radiotherapy; chemotherapy; Mucositis
MeSH Terms: conditions — Stomatitis; Ulcer; Mucositis | interventions — dexpanthenol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- normal saline (Experimental): mouth wash of normal saline ,three times a day, 10 cc each time
  Interventions: Drug: Dexpanthenol

INTERVENTIONS:
Drug: Dexpanthenol — 5% dexpanthenol Mouth wash , three times a day, 10 cc each time
  Other Names: Physiologic serum

SUMMARY:
Oral mucositis can be a significant problem for cancer patients. It is typically associated with pain and increased risk of infection and can lead to impaired nutritional status and inadequate hydration.it can be seen in the patient population receiving high-dose head and neck radiation therapy (85%-100%). Topical dexpanthenol acts like a moisturizer, improving stratum corneum hydration, reducing transepidermal water loss and maintaining skin softness and elasticity. The stimulation of epithelization, granulation and mitigation of itching were the most prominent effects of formulations containing dexpanthenol. The investigators suppose that dexpanthenol mouth wash may improve oral mucositis.

DETAILED DESCRIPTION:
Patients will be given a bottle of 5% Dexpanthenol mouthwash and they are asked to rinse 10 ml of it three times a day. At the onset of mucositis and then for 4 subsequent weeks they will be examined to evaluate the condition of their oral mucosa.By the advent of mucositis stage 4 ,at any time during the 4 weeks of study,the patient would be out.if any patient shows allergic reaction to dexpanthenol,he/she would be out of study too.

ELIGIBILITY:
Inclusion Criteria:

1. without any systemic disease
2. estimated survival of at least 6 months
3. without any mental disorders
4. grade 1 to 3 WHO mucositis

Exclusion Criteria:

1. development of grade 4 WHO mucositis
2. Brachytherapy
3. allergy to the drug
4. dissatisfaction of the patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
reduction of intensity of mucositis | first week (week one)
  measuring of the intensity of mucositis by visual examination and asking the patient about pain and discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Fahimeh Anbari, resident, Principal Investigator — dental faculty of shaheed Beheshti medical university
Locations (1):
- ShaheedBeheshti medical university, Tehran, Iran